CLINICAL TRIAL: NCT05207852
Title: Clinical Pharmacology of Dexamethasone in Pregnant Women With Preterm Labor
Status: Recruiting | Type: Observational
Sponsor: Dongyang Liu (Other)
Responsible Party: Sponsor-Investigator, Dongyang Liu, Vice director of Drug Clinical Trial Center, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: DCTC-IIR202108
Record Dates: First submitted 2021-12-13; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Distress Syndrome of Newborn; Threatened Premature Labor, Antepartum
Keywords: Dexamethasone; Pregnancy; Preterm; Quantitative pharmacology; P-glycoprotein
MeSH Terms: conditions — Pulmonary Atelectasis; Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood; placenta
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- 0.5 h group: Blood samples were taken 0.5 h after dexamethasone administration
- 2 h group: Blood samples were taken 2 h after dexamethasone administration
- 4 h group: Blood samples were taken 4 h after dexamethasone administration
- 6 h group: Blood samples were taken 6 h after dexamethasone administration
- 12 h group: Blood samples were taken 12 h after dexamethasone administration
- 24 h group: Blood samples were taken 24 h after dexamethasone administration
- 36 h group: Blood samples were taken 36 h after dexamethasone administration
- 48 h group: Blood samples were taken 48 h after dexamethasone administration

SUMMARY:
This study through to the pregnant woman blood concentrations of dexamethasone therapy after research, explore the pharmacokinetic data of dexamethasone in pregnant women, Chinese pregnant women dexamethasone pharmacokinetic model, provide a reference for the clinical use of dexamethasone dose, through the biomarkers of dexamethasone to promote fetal lung maturity and other metabolomics, It provides the basis for the effectiveness and safety study of dexamethasone.

DETAILED DESCRIPTION:
This study was a single-center, open clinical study. Maternal blood, feces, umbilical venous blood, and placental tissue were collected from GW24-36 Chinese women with preterm labor treated with dexamethasone, excluding placental abruption, severe intrauterine bleeding, or women who met the exclusion criteria. The determination and implementation of dexamethasone treatment by clinicians are executed according to the guidelines, the sample collected in addition to collecting feces and an active medication before an initiative to collect blood after medication, the other is to pregnant women normal diagnosis and treatment after operation opportunity or placental blood collection way, this study does not interfere with the normal of maternal pregnancy, production, and diagnosis and treatment process. A total of 288 Chinese pregnant women with preterm preterm birth who required dexamethasone treatment were randomly divided into eight groups with 36 participants in each group. At admission, blood was retained for each group after biochemical or routine blood test and blood was abandoned once (2 mL). After that, subjects were treated with DEX (5 mg intramuscularization, Q12h, for 2 days, if there was still no delivery 7 days after the first drug administration, another course of treatment or treatment as prescribed by the doctor). During the study period, do not take any food or drugs (such as coffee, alcohol, hypoglycemic drugs and other drugs used with caution or prohibited by pregnant women) that may affect the safety of the fetus. 2 mL of venous blood was collected from each group at 0.5 h, 2 h, 4 h, 6 h, 12 h, 24 h, 36 h, 48 h after the first administration. Blood biochemical or blood routine waste blood at the last prenatal examination was collected in each group, and umbilical venous blood was collected postpartum. Placenta samples were collected postpartum. All samples will be tested for dexamethasone and its metabolite concentrations, pharmacodynamics and safety indicators, hormones and metabolomics. Neonatal development was evaluated by PEABODY score and Bailey Scale at 6 and 24 months postnatal.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-40 (inclusive);
* Body mass Index (BMI) 18.5-27.9kg /m2 (inclusive)
* Single and twin pregnancy;
* Premature delivery at 24-36 weeks;
* No antibiotics, prebiotics or probiotics were used one month before feces collection (such as Bifidobacterium triplex live powder, Lactobacillus acidophilus tablet, compound Lactobacillus acidophilus tablet, Bacillus subtilis diplex live intestinal capsule, etc.);
* Preeclampsia patients accounted for about 1/10 of each group;
* Use dexamethasone I.M. 5mg Q12h regimen (or other dexamethasone administration regimen) to promote fetal lung maturation.

Exclusion Criteria:

* Ectopic pregnancy;
* Suffering from diabetes, fetal distress, serious infectious diseases (such as sepsis, septic shock), fever;
* Those who have taken glucocorticoid drugs within 2 weeks before joining the clinical trial;
* Those who took clindamycin during the study period;
* Congenital fetal malformation or fetal hypoxia in early pregnancy;
* Convulsive patients;
* HIV/HCV/ HEPATITIS A, drug abuse history;
* Suffering from chorioamnitis, endometritis;
* Placental abruption, severe intrauterine bleeding;
* Pregnant women whose cervical dilation is greater than or equal to 4 cm or whose cervical length is less than or equal to 20 mm by ultrasound examination;
* Pregnant women who took food or drugs during the study that might affect the safety of the fetus;
* Pregnant women participating in other clinical trials.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: 288 Chinese pregnant women with preterm prematurity requiring dexamethasone treatment.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory distress syndrome | At birth
  Whether respiratory distress syndrome occurs
hypoglycemia | Within 24 hours of birth
  Record fetal blood glucose (hypoglycemia within 1 hour, 3 hours, 6 hours, 24 hours after birth)
PEABODY | Six months
  Evaluate the mental and physical development of the newborn, including 2, 1 and 0, of which 2 is the best and 0 is the worst.
PEABODY | Two years
  Evaluate the mental and physical development of the newborn, including 2, 1 and 0, of which 2 is the best and 0 is the worst.
BayleyScales of Infant and Toddler Development | Six months
  Evaluate the mental and physical development of the newborn. Each infant's score on the Mental and motor scales was converted by age group into a standard score with an average of 100 and a standard deviation of 16, The Mental Development Index and Psychomotor Development Index were calculated.
BayleyScales of Infant and Toddler Development | Two years
  Evaluate the mental and physical development of the newborn. Each infant's score on the Mental and motor scales was converted by age group into a standard score with an average of 100 and a standard deviation of 16, The Mental Development Index and Psychomotor Development Index were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Dongyang, Principal Investigator — Drug Clinical Trial Center
Locations (1):
- Dongyang Liu, Beijing, China

IPD SHARING:
Plan to Share IPD: No